CLINICAL TRIAL: NCT06715267
Title: Children, Adolescents and Young Adults with Myeloproliferative Neoplasia: Study of Clinico-biological Characteristics and Complications
Brief Title: Children, Adolescents and Young Adults with Myeloproliferative Neoplasia: Study of Clinico-biological Characteristics and Complications (VYP)
Acronym: VYP
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC23.0018 - VYP
Record Dates: First submitted 2024-08-20; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Myeloproliferative Neoplasm
MeSH Terms: conditions — Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The creation of a national database will provide access to solid data on the diagnosis of myeloproliferative neoplasia for patients under 30, giving a true picture of their care. It will also make it possible to identify the biological samples (histological and molecular) available in routine laboratories, enabling teams of researchers and anatomopathologists to (re)perform certain analyses to re-evaluate diagnoses and search for hitherto unknown molecular prognostic factors.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with non-LMC MPN before the age of 30 (PV or TE or MFP or PreMF) according to the 2016 WHO criteria.
* Signature of the consent form for participation in the FIMBANK project.
* Agreement to participate in the VYP study.
* Patient of legal age at the time of inclusion in VYP.
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Refusal to participate by patients of full age
* Patient under legal protection (guardianship, curatorship, etc.)

Ages: 0 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients diagnosed with non-LMC myeloproliferative neoplasm before age 30 (Polycythemia vera, essential thrombocythemia, primary myelofibrosis, prefibrotic myelofibrosis).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2038-04-01 (Estimated); Study Completion 2038-04-01 (Estimated)

PRIMARY OUTCOMES:
Describe the epidemiological characteristics of the study population | at enrollment
  Description of MPN subtypes according to age
Describe the mutational landscape of these MPNs | at enrollment
  Rate of mutations JAK2/CALR/MPL

SECONDARY OUTCOMES:
Describe the classical MPN (Myeloproliferative neoplasia) outcomes-1 | At 10 years
  Incidence of thrombosis
Describe the classical MPN outcomes-2 | At 10 years
  Incidence of myelofibrosis
Describe the classical MPN outcomes-3 | At 10 years
  Incidence of MDS/AML

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.